CLINICAL TRIAL: NCT01839318
Title: Subjective Comparison of Pre-Lens Tear Film Stability With Daily Disposable Contact Lenses Using Ring Mire Projection
Brief Title: Subjective Comparison of Pre-Lens Tear Film Stability With Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A01336
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-05

CONDITIONS: Myopia; Hyperopia; Refractive Error
Keywords: Soft contact lenses; Daily disposable contact lenses; Tear Film Break Up Time; Contact lens wettability
MeSH Terms: conditions — Myopia; Hyperopia; Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DAILIES AquaComfort Plus (Experimental): Nelfilcon A contact lenses worn first, followed by etafilcon A and omafilcon A in randomized order. Each product worn for 1 day, 12 hours.
  Interventions: Device: Nelfilcon A contact lenses
- 1-DAY ACUVUE MOIST (Active Comparator): Etafilcon A contact lenses worn first, followed by nelfilcon A and omafilcon A in randomized order. Each product worn for 1 day, 12 hours.
  Interventions: Device: Etafilcon A contact lenses
- Proclear 1 day (Active Comparator): Omafilcon A contact lenses worn first, followed by etafilcon A and nelfilcon A in randomized order. Each product worn for 1 day, 12 hours.
  Interventions: Device: Omafilcon A contact lenses

INTERVENTIONS:
Device: Nelfilcon A contact lenses
  Other Names: DAILIES® AquaComfort Plus®
  Arms: DAILIES AquaComfort Plus
Device: Omafilcon A contact lenses
  Other Names: Proclear® 1 day
  Arms: Proclear 1 day
Device: Etafilcon A contact lenses
  Other Names: 1-DAY ACUVUE® MOIST®
  Arms: 1-DAY ACUVUE MOIST

SUMMARY:
The purpose of this study was to compare three CE-marked daily disposable contact lenses for tear film stability as measured by pre-lens non-invasive keratograph break up time (PL NIK-BUT). Secondarily, contact lens surface wettability was assessed.

DETAILED DESCRIPTION:
Each participant wore 3 brands of contact lenses in a randomized, cross-over fashion, with a washout phase of at least 1 night between brands.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent.
* Adapted soft contact lens wearer.
* Willing to wear contact lenses up to 12 hours and attend all study visits.
* Vision correctable to 0.1 (logMAR) or better in each eye at distance with pre-study lenses at Visit 1.
* Contact lens prescription within the power range specified in the protocol.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any ocular infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear.
* Any use of systemic or ocular medications that would contraindicate contact lens wear.
* Any ocular finding observed during the Visit 1 examination that would contraindicate contact lens wear.
* Monocular (only 1 eye with functional vision) or fit with only 1 lens.
* History of herpetic keratitis, ocular surgery, or irregular cornea.
* Known pregnancy.
* Unstable tear film with a NIK-BUT value below 13 seconds in either eye without lenses.
* Participation in any clinical study within 30 days of Visit 1.
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Lemp, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in Germany.
Pre-assignment Details: Of the 30 enrolled, 2 participants discontinued before product was dispensed. This reporting group includes all participants exposed to the study product (28). In this 3-treatment, 6-sequence crossover study, each participant received all 3 products in randomized order and used 1 product at a time for a duration of 12 hours.
Groups:
- Sequence 1: Omafilcon A contact lenses worn first, followed by nelfilcon A contact lenses worn second, then etafilcon A contact lenses worn last. Each product worn for 1 day, 12 hours.
- Sequence 2: Omafilcon A contact lenses worn first, followed by etafilcon A contact lenses worn second, then nelfilcon A contact lenses worn last. Each product worn for 1 day, 12 hours.
- Sequence 3: Nelfilcon A contact lenses worn first, followed by etafilcon A contact lenses worn second, then omafilcon A contact lenses worn last. Each product worn for 1 day, 12 hours.
- Sequence 4: Nelfilcon A contact lenses worn first, followed by omafilcon A contact lenses worn second, then etafilcon A contact lenses worn last. Each product worn for 1 day, 12 hours.
- Sequence 5: Etafilcon A contact lenses worn first, followed by omafilcon A contact lenses worn second, then nelfilcon A contact lenses worn last. Each product worn for 1 day, 12 hours.
- Sequence 6: Etafilcon A contact lenses worn first, followed by nelfilcon A contact lenses worn second, then omafilcon A contact lenses worn last. Each product worn for 1 day, 12 hours.
Period: Period 1, First Day of Wear
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 4 | 5 | 6 | 7 | 2
Completed | 4 | 4 | 5 | 6 | 7 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2, Second Day of Wear
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 4 | 5 | 6 | 7 | 2
Completed | 4 | 4 | 5 | 6 | 7 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3, Third Day of Wear
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 4 | 5 | 6 | 7 | 2
Completed | 4 | 4 | 5 | 6 | 7 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants who were exposed to a study product.
Groups:
- Overall: Nelfilcon A contact lenses, etafilcon A contact lenses, and omafilcon A contact lenses worn in a cross-over assignment.
Arm/Group | Overall
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.96 (3.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Pre-Lens Non-Invasive Keratograph Break Up Time (PL NIK-BUT) at 8 Hours
Description: The pre-lens tear film is the layer of tears located on top of the contact lens (i.e., between the eye lid and the contact lens). The time required for a dry spot to appear on the corneal surface after blinking is referred to as the tear film break-up time. Circular images were projected onto the contact lens using an Oculus Keratograph 5 and the tear film reflection was observed. PL NIK-BUT was recorded at the first sign of distortion. A longer tear film break-up time indicates a more stable tear film. One eye (right eye) contributed to the mean.
Time Frame: Hour 8
Population: This analysis population includes all participants exposed to the study product with reportable values.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- DAILIES AquaComfort Plus: Nelfilcon A contact lenses worn in a randomized order for 1 day, 12 hours
- 1-DAY ACUVUE MOIST: Etafilcon A contact lenses worn in a randomized order for 1 day, 12 hours
- Proclear 1 Day: Omafilcon A contact lenses worn in a randomized order for 1 day, 12 hours
Arm/Group | DAILIES AquaComfort Plus | 1-DAY ACUVUE MOIST | Proclear 1 Day
Number analyzed (Participants) | 27 | 26 | 27
seconds | 5.28 (5.71) | 3.46 (4.52) | 4.93 (6.34)

2. Secondary Outcome: Total Wettability Score
Description: The investigator graded lens wettability by corneal region using a scale from 0 (fully wettable) to 3 (clearly visible ring distortions in more than 1/3 of ring reflection zone). The total wettability score per eye was calculated by averaging the grade of each of the 5 corneal regions (central, superior, nasal, inferior, and temporal). One eye (right eye) contributed to the mean.
Time Frame: Hour 8
Population: This analysis population includes all participants exposed to the study product with reportable values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DAILIES AquaComfort Plus | 1-DAY ACUVUE MOIST | Proclear 1 Day
Number analyzed (Participants) | 27 | 26 | 27
units on a scale
  5 seconds post blink | 0.74 (0.93) | 0.83 (0.87) | 0.84 (0.96)
  10 seconds post blink | 1.25 (1.15) | 1.20 (1.14) | 1.42 (1.2)
  15 seconds post blink | 1.58 (1.2) | 1.54 (1.21) | 1.66 (1.19)
  20 seconds post blink | 1.69 (1.21) | 1.78 (1.22) | 1.89 (1.18)
  25 seconds post blink | 1.79 (1.18) | 1.94 (1.19) | 2.03 (1.17)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (2 months). This analysis group includes all enrolled participants.
Description: An AE is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device.
Arm/Group | DAILIES AquaComfort Plus | 1-DAY ACUVUE MOIST | Proclear 1 Day
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.